CLINICAL TRIAL: NCT04977089
Title: Study of Lipid Profile of Patients With Chronic Coronary Syndromes at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Farrag, resident doctor at internal medicine department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-07-01
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Heart Disease; Dyslipidemias
MeSH Terms: conditions — Myocardial Ischemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic heart disease patients .: Study of lipid profile of patients with chronic coronary syndromes who recieve drugs of anti hyperlipidemia at the cardiology clinic of sohag university hospital.
  Interventions: Diagnostic Test: lipid profile test .

INTERVENTIONS:
Diagnostic Test: lipid profile test . — Assesment of lipid profile of patients (cholesterol level ,TG ,VLDL )

SUMMARY:
Chronic coronary syndrome (CCS) is a newly described classification devised by the European Society of Cardiology (ESC) 2019 to replace the term "Stable Coronary Artery Disease (CAD).

The main reason for effecting the change is the term is thought to better describe the disease process and encompass a wider spectrum of clinical, pharmacological, and pathophysiological entities.

Using this new term, the disease atherosclerosis manifests as CAD is categorized into Acute Coronary Syndrome (ACS) and CCS.

The main focus of introducing the concept of CCS is on the fact that CAD is a continuous phenomenon involving intravascular plaque aggregation and progression which has different evolutionary phases.

Dyslipidemia is recognized as a prominent risk factor for cardiovascular (CV) disease.

It is characterized by an elevation of serum total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), or triglycerides (TG) and reduced serum high-density lipoprotein cholesterol (HDL-C) concentration .

Genetically determined and metabolically induced disturbances in lipid metabolism, as manifested in several types of dyslipidemia, have been shown to be causally related to the development of coronary artery disease (CAD).

A diversity of clinical and angiographic studies has been made to evaluate the linkage between plasma lipid-control therapy in the development of recurrent cardiovascular events.

Independent predictors of recurrent CVD events or death include age, smoking, hypertension (HTN), dyslipidemia, diabetes mellitus, chronic kidney disease, and the underutilization of medications recommended by current treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients have chronic coronary disease at Sohag University hospital who recieve drugs of anti hyperlipidemia .

Exclusion Criteria:

* Patients with first attack of acute coronary syndrome .
* Young patients <18 years .
* Old patients >65 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: I examine cross sectional study which classify 100 patients with chronic coronary syndrome into:
  two main groups :
  * patient on statin therapy.
  * patient not on statin therapy. _And determine if patints in sohag university hospital could achive the target lipid profile level of their group according to 2019 ESC/EAS Guidelines for the management of dyslipidaemia.
  I classify 100 patients with chronic coronary syndrome into:
  two main groups :
  * patient on statin therapy.
  * patient not on statin therapy. _And determine if patints in sohag university hospital could achive the target lipid profile level of their group according to 2019 ESC/EAS Guidelines for the management of dyslipidaemia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Dyslipidemia in chronic coronary syndrome | one year
  Pattern of dyslipidemia among patients with chronic coronary syndromes at sohag university hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Darroudi S, Saberi-Karimian M, Tayefi M, Arekhi S, Motamedzadeh Torghabeh A, Seyedzadeh Sani SMR, Moohebati M, Heidari-Bakavoli A, Ebrahimi M, Azarpajouh MR, Safarian M, A Ferns G, Esmaeili H, Parizadeh MR, Mokhber N, Mahdizadeh A, Mahmoudi AA, Sahebkar AH, Ghayour-Mobarhan M. Prevalence of combined and noncombined dyslipidemia in an Iranian population. J Clin Lab Anal. 2018 Oct;32(8):e22579. doi: 10.1002/jcla.22579. Epub 2018 Jun 21. PMID 29926995
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Mortensen MB, Falk E, Li D, Nasir K, Blaha MJ, Sandfort V, Rodriguez CJ, Ouyang P, Budoff M. Statin Trials, Cardiovascular Events, and Coronary Artery Calcification: Implications for a Trial-Based Approach to Statin Therapy in MESA. JACC Cardiovasc Imaging. 2018 Feb;11(2 Pt 1):221-230. doi: 10.1016/j.jcmg.2017.01.029. Epub 2017 Jul 25. PMID 28624395